CLINICAL TRIAL: NCT04251299
Title: Southwest Harvest for Health: A Mentored Vegetable Gardening Intervention for Cancer Survivors in New Mexico
Brief Title: Southwest Harvest for Health Vegetable Gardening Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of New Mexico (Other)
Collaborators: University of New Mexico Cancer Center (Other); New Mexico State University (Other)
Responsible Party: Principal Investigator, Cindy Blair, PhD, MPH, Assistant Professor, University of New Mexico
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: INST UNM 1905
Record Dates: First submitted 2020-01-24; First posted 2020-01-31 (Actual); Results first posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Cancer Survivor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Arm (Experimental): All participants will receive the 10-month mentored, vegetable gardening intervention
  Interventions: Behavioral: home-based, mentored vegetable gardening program

INTERVENTIONS:
Behavioral: home-based, mentored vegetable gardening program — The mentored vegetable gardening program pairs each participant with a certified Master Gardener. The participant/Master Gardener dyads work together to plan, plant and tend to a vegetable garden at the participant's home throughout the year. Gardening supplies, plants and seeds are provided.

SUMMARY:
"Harvest for Health" is a home-based vegetable gardening intervention that pairs cancer survivors with certified master gardeners (MGs) from the Cooperative Extension System, the education and outreach arm of land-grant universities nationwide.

DETAILED DESCRIPTION:
Few lifestyle behavior change interventions have been successfully translated into practice. Addressing this research-to-practice gap is a significant research and public health priority. "Harvest for Health" is a home-based vegetable gardening intervention that pairs cancer survivors with certified Master Gardeners from the Cooperative Extension System. The parent study was started at the University of Alabama at Birmingham and is currently being conducted throughout the entire state of Alabama. Preliminary findings suggest that this intervention increases vegetable consumption and physical activity, and improves physical functioning and health-related quality of life. We propose a feasibility study to adapt this promising program to the multi-cultural population of cancer survivors and for the local context (physical, social, and cultural environment) of New Mexico. We will then implement the adapted program, "Southwest Harvest for Health" and evaluate feasibility, acceptability, and fidelity. The adaptation phase is a critical first step towards widespread dissemination, implementation, and scale-up of an evidence-based intervention.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 years or older
* Residing in Bernalillo or Sandoval County, New Mexico
* Diagnosed with an invasive cancer (any type)
* Completed primary treatment (surgery, radiation, chemotherapy)(note: endocrine therapy is allowed)
* Able to read, speak, and understand English (The future larger trial will include Spanish-Speaking participants)
* Not told by a physician to limit physical activity and no pre-existing medical condition(s) that would preclude home gardening, e.g., severe orthopedic conditions, hip or knee replacement surgery within 6 months), end-stage renal disease, paralysis, dementia, blindness, unstable angina, untreated stage 3 hypertension, or recent history of myocardial infarction, congestive heart failure, or pulmonary conditions that required oxygen or hospitalization within 6 months.
* Currently not adhering to the recommended number of fruit and vegetable servings per day (consuming fewer than 5 servings of vegetables and fruits/day and not meeting the recommended guidelines for moderate-to-vigorous physical activity (< 150 minutes/week)
* Reside in a location that can accommodate a 4' x 8' raised garden bed or 4 (29" x 14") garden containers, or adequate (at least 4 hours) of sunlight per day and have access to running water
* No existing or recent (within the past year) experience with vegetable gardening
* Able to participate in the 10-month intervention (all three seasonal gardens; from mid-February through early November 2020)

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-01-17 (Actual); Primary Completion 2020-12-20 (Actual); Study Completion 2020-12-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cindy K Blair, PhD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Distributed recruitment flyers in community locations, e.g., cancer survivor support groups, community centers. Also, oncologists, physicians, and nurse navigators referred patients (cancer survivors). Self-referrals.
  Note: Master Gardeners are not participants; they were not enrolled and consented, nor did they complete outcome assessments; instead, they are volunteers from the Extension Master Gardener Program who delivered the interention.
Period: Overall Study
Arm/Group | Single Arm
Started | 30 (30 cancer survivors were enrolled in the study.)
Completed | 30 (All cancer survivors enrolled received the mentored gardening intervention.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Only the cancer survivors enrolled in the study completed the baseline and post-intervention assessments. The Master Gardener mentors delivered the intervention.
Arm/Group | Single Arm
Number analyzed (Participants) | 30
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21
  Male | 9
Race/Ethnicity, Customized [Number; unit: participants]
  Non-Hispanic White | 22
  Hispanic White | 6
  Other | 2
Region of Enrollment [Number; unit: participants]
  United States | 30

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Intervention
Description: Ability to recruit 25 cancer survivors in 3 months, achieve 80% retention rates, 80% adherence to the intervention, and high acceptability of the program for both cancer survivors (participants) and Cooperative Extension Master Gardeners.
Time Frame: through study completion, an average of 9 months
Population: (1) Percentage of participants recruited within 3 months; (2) percentage of participants who completed the study; (3) percentage of participants adhering to twice monthly communication with Master Gardener mentor; (4) percentage rating their experience with the intervention as very good or excellent.
Measure: Number; unit: percentage of participants
Arm/Group | Single Arm
Number analyzed (Participants) | 30
percentage of participants
  Percentage recruited within 3 months | 100
  Percent retention (completed study) | 100
  Percentage adherence (twice monthly communication with mentor) | 89
  Percentage Satisfaction (very good or excellent) | 90

2. Secondary Outcome: Pre-post Change in Vegetable and Fruit Intake
Description: The number of daily servings of vegetables and fruits will be measured by the Eating at America's Table Screener (EATS) questionnaire; this 10-item NCI-developed questionnaire will be able to assess whether individuals increase by more than one serving of vegetables/fruits per day.
Time Frame: baseline to 9-months
Measure: Median (Inter-Quartile Range); unit: fruit & vegetable servings/day
Arm/Group | Single Arm
Number analyzed (Participants) | 30
fruit & vegetable servings/day | 1.2 [-0.4 to 2.2]

3. Secondary Outcome: Pre-post Change in Objectively Measured Physical Activity
Description: Physical activity will be objectively measured using the activPAL research grade monitor.
Time Frame: baseline to 9-months
Measure: Median (Inter-Quartile Range); unit: minutes per day
Arm/Group | Single Arm
Number analyzed (Participants) | 30
minutes per day
  light-intensity physical activity | -1.1 [-10.6 to 3.4]
  moderate-intensity physical activity | -4.2 [-13.8 to 3.7]

4. Secondary Outcome: Pre-post Change in Sleep Quality
Description: Self-reported sleep quality will be assessed using the PROMIS 8-item questionnaires for sleep impairment and sleep disturbance. Raw scores range from 8 to 40; higher scores indicate worse sleep quality; T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean.
Time Frame: baseline to 9-months
Measure: Median (Inter-Quartile Range); unit: change in points
Arm/Group | Single Arm
Number analyzed (Participants) | 30
change in points
  Sleep disturbance | -0.4 [-1.7 to 2.4]
  Sleep impairment | -0.2 [-6.0 to 5.1]

5. Secondary Outcome: Pre-post Change in Physical Function
Description: Self-reported physical function will be assessed using the 8-item physical function scale. Raw scores range from 8 to 40; higher scores indicate better physical function; T-score rescales the raw score into a standardized score with a mean of 50 and a standard deviation (SD) of 10. Therefore, a person with a T-score of 40 is one SD below the mean.
Time Frame: baseline to 9-months
Measure: Median (Inter-Quartile Range); unit: change in points
Arm/Group | Single Arm
Number analyzed (Participants) | 30
change in points | 0.0 [-7.0 to 4.3]

6. Secondary Outcome: Pre-post Change in Physical Performance
Description: Physical performance will be objectively measured using the Rikli & Jones Senior Fitness Battery.
Time Frame: baseline to 9-months
Population: Due to the COVID-19 pandemic, the in-person assessment of physical performance was dropped. Studies at the University of New Mexico were not allowed to conduct in-person assessments in 2020 after the pandemic was declared. Therefore, no post-intervention data on physical performance was collected (for any participant), and it is not possible to calculate change in physical performance. Only baseline physical performance data was collected.
Arm/Group | Single Arm
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 9 months
Groups:
- Single Arm: All participants (cancer survivors) will receive the 10-month mentored, vegetable gardening intervention home-based, mentored vegetable gardening program: The mentored vegetable gardening program pairs each participant with a certified Master Gardener. The participant/Master Gardener dyads work together to plan, plant and tend to a vegetable garden at the participant's home throughout the year. Gardening supplies, plants and seeds are provided. Note: Data are not collected for Master Gardeners who deliver the intervention; neither baseline data, post-intervention data, nor adverse events are collected/recorded for Master Gardeners.
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/30
Serious Adverse Events (participants affected / at risk) | 0/30
Other Adverse Events (participants affected / at risk) | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2020-11-01): https://cdn.clinicaltrials.gov/large-docs/99/NCT04251299/Prot_SAP_ICF_000.pdf